CLINICAL TRIAL: NCT03506035
Title: Alloimmune Model in Rheumatoid Arthritis. Alloimmune Response to Citrullinated Shared Epitope Sequence in Patients With Rheumatoid Arthritis.Alloimmune Response to Citrullinated Shared Epitope Sequence in Patients With Rheumatoid Arthritis
Brief Title: Alloimmune Response to Citrullinated Shared Epitope Sequence in Patients With Rheumatoid Arthritis
Acronym: ABSEC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Eduard Graell-Martin, MD. PhD, Corporacion Parc Tauli
Other Study IDs: CIR2017/011
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Shared epitope; HLA-DRB1; Citrullinated peptides; Autoantibodies
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rheumatoid arthritis: Patients who meet the criteria of the 1987 ACR
  Interventions: Diagnostic Test: Research new biomarker for RA
- Arthritis not Rheumatoid arthritis: Patients with psoriatic arthritis, peripheric spondyloarthropathies and connective tissue diseases.
  Interventions: Diagnostic Test: Research new biomarker for RA
- Healthy controls: From health blood donors
  Interventions: Diagnostic Test: Research new biomarker for RA

INTERVENTIONS:
Diagnostic Test: Research new biomarker for RA — Analyze T and B cell response against new citrullinated peptides

SUMMARY:
Rheumatoid arthritis (RA) is an autoimmune and sistemic disease,characterized by joint sinovitis and the production of autoantibodies (Ab). The Ab against citrullinated peptides (ACPA) are the most specific (92-98%), and high sensitivity (75-81%) and they are of prognostic value. ACPA are already in the beginning of the disease in most cases, having been found years before its onset. Recent studies have suggested that ACPA may have a role in perpetuating inflammation, in the generation of bone erosions and in pain in RA.

Citrullination is a post-translational modification mediated by the PAD, which transforms an arginine into a citrulline. In vivo, this enzyme acts in proinflammatory environments. Despite being widely studied, none of the natural citrullinated substrates have been shown to be the triggering and/or perpetuating factor in the response of B cells in RA, understanding this response as the production of ACPA. In fact, the most specific and sensitive commercial test for the detection of ACPA uses synthetic peptides protected by a patent.

In the other hand, the genetic factor that most increases susceptibility to develop RA is a shared sequence of aminoacids (QKRAA, QRRAA i RRRAA), in the HLA-DRB1 gene, known as the shared epitope (SE). Also, SE, confers prognostic value, and is associated with the presence of ACPA. These SE sequences contain arginines (R), which are susceptible to be citrullinated by the PAD enzyme.

We propose the hypothesis that citrullinated SE act as an antigen capable of activating the inflammatory response mediated by B and T cells in RA. The recognition of an HLA as a foreign one, would originate an answer of alloimmune type, not valued to date.

The objective of the study is to test the immune response mediated by B cells and T cells, in cases and control samples, through an in vitro model that confronts them with peptides containing the citrullinated-SE sequence. In addition, we will evaluate the association between these results with the clinical features of cases (RA included in the study). Their role as a biomarker, as well as their potential to improve the tests currently available to detect ACPA will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA who meet 1987 ACR criteria Patients with arthritis no RA

Exclusion Criteria:

* Having an intellectual disability that allows understanding the informed consent to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from rheumatology outpatients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
T cell response | 2 years
  Proliferation against new citrullinated peptides
B cell response | 2 years
  Detection antibodies against new citrullinated peptides

SECONDARY OUTCOMES:
HLA-DRB1 | 2 years
  Typing HLA-DRB1
Rheumatic factor | 2 years
  Turbidimetric assay
Anti-Citrullinated Peptides Antibodies | 2 years
  ELISA assay

IPD SHARING:
Plan to Share IPD: Undecided